CLINICAL TRIAL: NCT03907280
Title: Absolute Bioavailability of BI 1265162 Following Oral and Inhaled Administration in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Three-period, Three-sequence Crossover Study Followed by a Fixed Treatment)
Brief Title: A Study in Healthy Men That Tests if Taking BI 1265162 by Mouth, Intravenously, or Inhaled Influences the Amount of BI 1265162 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1399-0014; 2018-002689-38 (EudraCT Number)
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1-T2-R-T3 (Experimental)
  Interventions: Drug: BI 1265162 (T1); Drug: BI 1265162 (T2); Drug: BI 1265162 (R); Drug: BI 1265162 (T3)
- R-T1-T2-T3 (Experimental)
  Interventions: Drug: BI 1265162 (T1); Drug: BI 1265162 (T2); Drug: BI 1265162 (R); Drug: BI 1265162 (T3)
- T2-R-T1-T3 (Experimental)
  Interventions: Drug: BI 1265162 (T1); Drug: BI 1265162 (T2); Drug: BI 1265162 (R); Drug: BI 1265162 (T3)

INTERVENTIONS:
Drug: BI 1265162 (T1) — oral solution
Drug: BI 1265162 (T2) — Solution for inhalation
Drug: BI 1265162 (R) — concentrate for i.v. solution
Drug: BI 1265162 (T3) — Solution for inhalation

SUMMARY:
The main objective of this trial is to investigate the absolute bioavailability of BI 1265162 following administration of oral solution and inhaled (with and without charcoal) via Respimat.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* The subject has a diagnosis history of pulmonary hyperreactivity
* A history of chronic kidney disease
* Cannot use Respimat® appropriately

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Mackie A, Rascher J, Schmid M, Endriss V, Brand T, Seibold W. First clinical trials of the inhaled epithelial sodium channel inhibitor BI 1265162 in healthy volunteers. ERJ Open Res. 2021 Feb 1;7(1):00447-2020. doi: 10.1183/23120541.00447-2020. eCollection 2021 Jan. PMID 33569494
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as a randomized, open-label, 3-way crossover trial followed by a fixed treatment in healthy male subjects in order to compare BI 1265162 given as oral solution (T1) and BI 1265162 inhaled via Respimat® with activated charcoal (T2) and without activated charcoal (fixed treatment, T3) compared with BI 1265162 given intravenously (R).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- (T1-T2-R-T3) Treatment Sequence; (R-T1-T2-T3) Treatment Sequence; (T2-R-T1-T3) Treatment Sequence: In this randomized, 3-way crossover trial followed by a fixed treatment participants were randomized to one of 3 possible treatment sequences. Treatments administered were 1.25 milligram (mg) of BI 1265162 as oral solution (5 milliliter (mL) of 0.25 mg/mL) administered orally with 240 mL of water after an overnight fast of at least 8 hours (h) (Test treatment 1, T1), 200 microgram (μg) of BI 1265162 as solution for inhalation (2 actuations of 100 μg) inhaled by Respimat® after an overnight fast of at least 8 h in combination with activated charcoal (Test treatment 2, T2) and without activated charcoal (Fixed treatment, Test treatment 3, T3), 50 μg of BI 1265162 concentrate for infusion (2 mL of 25 μg/mL) administered intravenously over 1 h after an overnight fast of at least 8 h (Reference treatment, R). Each treatment was administered as a single dose and a washout period of at least 6 days was adhered to between drug administrations.
Period: Treatment Period 1 + Washout Period 1
Arm/Group | (T1-T2-R-T3) Treatment Sequence | (R-T1-T2-T3) Treatment Sequence | (T2-R-T1-T3) Treatment Sequence
Started (= Randomized to treatment sequence) | 4 | 4 | 4
Treated With BI 1265162 | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Treatment Period 2 + Washout Period 2
Arm/Group | (T1-T2-R-T3) Treatment Sequence | (R-T1-T2-T3) Treatment Sequence | (T2-R-T1-T3) Treatment Sequence
Started (= Randomized to treatment sequence) | 4 | 4 | 4
Treated With BI 1265162 | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Treatment Period 3 + Washout Period 3
Arm/Group | (T1-T2-R-T3) Treatment Sequence | (R-T1-T2-T3) Treatment Sequence | (T2-R-T1-T3) Treatment Sequence
Started (= Randomized to treatment sequence) | 4 | 4 | 4
Treated With BI 1265162 | 4 | 3 | 4
Completed | 4 | 3 | 4
Not Completed | 0 | 1 | 0
Not completed — Not treated with BI 1265162 because of Serious Adverse Event in Treatment Period 2 | 0 | 1 | 0
Period: Treatment Period 4: Fixed Treatment T3
Arm/Group | (T1-T2-R-T3) Treatment Sequence | (R-T1-T2-T3) Treatment Sequence | (T2-R-T1-T3) Treatment Sequence
Started (= Randomized to treatment sequence) | 4 | 4 | 4
Treated With BI 1265162 | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All participants who were randomized and treated with at least 1 dose of any trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | (T1-T2-R-T3) Treatment Sequence | (R-T1-T2-T3) Treatment Sequence | (T2-R-T1-T3) Treatment Sequence | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.9) | 41.3 (7.9) | 39.8 (10.2) | 36.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1265162 in Plasma Over the Time Interval From 0 Extrapolated to Infinity, Dose-normalized, (AUC0-∞, Norm)
Description: Area under the concentration-time curve of BI 1265162 in plasma over the time interval from 0 extrapolated to infinity, dose-normalized to 1 µg BI 1265162, (AUC0-∞, norm).
  Time frame for treatment T1:
  Within 3 hours before and 30 and 45 minutes, 1, 2, 3, 4, 6, 8, 12 and 24 hours following administration of the trial drug.
  Time frame for treatment T2 and T3:
  Within 3 hours before and 2, 5, 10, 15 and 40 minutes, 1, 2, 4, 8, 10, 12 and 24 hours following administration of the trial drug.
  Time frame for treatment R:
  Within 3 hours (h) before and 5, 30 and 59 minutes (min), 1 h 5 min, 1 h 10 min, 1 h 20 min, 1 h 40 min, 2, 2 h 30 min, 3, 3 h 30 min, 4, 5, 7, 9, 11, 13 and 24 hours following administration of the trial drug.
Time Frame: Up to 24 hours following administration of the trial drug, see detailed time frame in the endpoint description.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): All participants who were randomized and treated with at least 1 dose of any trial drug and who provided at least 1 PK endpoint being defined as primary or further and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: ((hour * millimole) / liter) / kilogram
Groups:
- BI 1265162 as Infusion (R): 50 microgram (μg) of BI 1265162 concentrate for infusion (2 milliliter (mL) of 25 μg/mL) administered intravenously over 1 hour after an overnight fast of at least 8 hours (Reference treatment, R).
- BI 1265162 as Oral Solution (T1): 1.25 milligram (mg) of BI 1265162 as oral solution (5 milliliter (mL) of 0.25 mg/mL) administered orally with 240 mL of water after an overnight fast of at least 8 hours (Test treatment 1, T1).
- BI 1265162 for Inhalation With Activated Charcoal (T2): 200 microgram (μg) of BI 1265162 as solution for inhalation (2 actuations of 100 μg) inhaled by Respimat® after an overnight fast of at least 8 hours in combination with activated charcoal (Test treatment 2, T2).
- BI 1265162 for Inhalation Without Activated Charcoal (T3): 200 microgram (μg) of BI 1265162 as solution for inhalation (2 actuations of 100 μg) inhaled by Respimat® after an overnight fast of at least 8 hours without activated charcoal (Fixed treatment, Test treatment 3, T3).
Arm/Group | BI 1265162 as Infusion (R) | BI 1265162 as Oral Solution (T1) | BI 1265162 for Inhalation With Activated Charcoal (T2) | BI 1265162 for Inhalation Without Activated Charcoal (T3)
Number analyzed (Participants) | 12 | 12 | 11 | 12
((hour * millimole) / liter) / kilogram | 44.63 (NA) — Standard Error is geometric Standard Error (gSE) = 1.11. | 0.22 (NA) — Standard Error is geometric Standard Error (gSE) = 1.11. | 17.97 (NA) — Standard Error is geometric Standard Error (gSE) = 1.11. | 17.96 (NA) — Standard Error is geometric Standard Error (gSE) = 1.11.
Statistical Analysis 1: Comparison: BI 1265162 as Infusion (R) vs BI 1265162 as Oral Solution (T1); Exploratory trial, no formal hypotheses were tested. Analysis of variance (ANOVA) on the logarithmic scale including effects for treatment sequence ('fixed effect'), subjects nested within treatment sequences ('random effect'), and treatment ('fixed effect'); Test type: Other — Absolute bioavailability comparison; Mixed Models Analysis; Ratio of the geometric means (T1/R) [%] = 0.5, 90% CI 2-sided [0.39 to 0.63], Standard Error of Mean 1.15 — The standard error of the mean is actually the geometric standard error
Statistical Analysis 2: Comparison: BI 1265162 as Infusion (R) vs BI 1265162 for Inhalation With Activated Charcoal (T2); [analysis description as in outcome 1, analysis 1]; Test type: Other — Absolute bioavailability comparison; Mixed Models Analysis; Ratio of the geometric means (T2/R) [%] = 40.26, 90% CI 2-sided [31.68 to 51.15], Standard Error of Mean 1.15 — The standard error of the mean is actually the geometric standard error
Statistical Analysis 3: Comparison: BI 1265162 as Infusion (R) vs BI 1265162 for Inhalation Without Activated Charcoal (T3); [analysis description as in outcome 1, analysis 1]; Test type: Other — Absolute bioavailability comparison; Mixed Models Analysis; The standard error of the mean is actually the geometric standard error; Ratio of the geometric means (T3/R) [%] = 40.24, 90% CI 2-sided [31.86 to 50.83], Standard Error of Mean 1.15

ADVERSE EVENTS:
Time Frame: For Serious and Other Adverse Events: On-treatment period, that is, from administration of the respective formulation of BI 1265162 until the end of the residual effect period, up to 2 days. For All-Cause Mortality: Each on-treatment period + Follow-up period, i.e. up to 48 days.
Description: Treated set (TS): All participants who were randomized and treated with at least 1 dose of any trial drug.
Arm/Group | BI 1265162 as Infusion (R) | BI 1265162 as Oral Solution (T1) | BI 1265162 for Inhalation With Activated Charcoal (T2) | BI 1265162 for Inhalation Without Activated Charcoal (T3)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12 | 0/11 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1265162 as Infusion (R) (N=12) | BI 1265162 as Oral Solution (T1) (N=12) | BI 1265162 for Inhalation With Activated Charcoal (T2) (N=11) | BI 1265162 for Inhalation Without Activated Charcoal (T3) (N=12)
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1265162 as Infusion (R) (N=12) | BI 1265162 as Oral Solution (T1) (N=12) | BI 1265162 for Inhalation With Activated Charcoal (T2) (N=11) | BI 1265162 for Inhalation Without Activated Charcoal (T3) (N=12)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03907280/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03907280/SAP_001.pdf